CLINICAL TRIAL: NCT04076618
Title: Incorporating Nutrition, Vests, Education, and Strength Training in Bone Health (INVEST in Bone Health)
Acronym: INVEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB00058279
Record Dates: First submitted 2019-08-29; First posted 2019-09-03 (Actual); Results first posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-04

CONDITIONS: Weight Loss; Bone Health
Keywords: nutrition; vest
MeSH Terms: conditions — Weight Loss | interventions — Resistance Training; Weight Reduction Programs

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Weight Loss plus Vest (Experimental)
  Interventions: Device: Vest; Behavioral: weight loss program
- Weight Loss Plus Resistance Exercise Training (Active Comparator)
  Interventions: Behavioral: Resistance Exercise Training; Behavioral: weight loss program
- Weight Loss (Active Comparator)
  Interventions: Behavioral: weight loss program

INTERVENTIONS:
Device: Vest — Weighted Vest worn > or = 8 hours per day
  Arms: Weight Loss plus Vest
Behavioral: Resistance Exercise Training — Structured exercise training 3 days a week
  Arms: Weight Loss Plus Resistance Exercise Training
Behavioral: weight loss program — a 24-week intensive phase (with weekly dietary classes) followed by a 27-week transition phase (with biweekly dietary classes)

SUMMARY:
The main goal of the proposed study is to compare the effects of weight loss (WL) alone with WL plus weighted vest use or WL plus resistance exercise training (RT) on indicators of bone health and subsequent fracture risk.

DETAILED DESCRIPTION:
The study team proposes that a 12 month trial in 150 older (60-85 years) adults with obesity (Body mass index or BMI=30-40 kg/m2 OR 27.0-<30 kg/m² and one obesity-related risk factor) randomized to one of three interventions (n=50/group): WL alone (WL; caloric restriction targeting 10% WL); WL plus weighted vest use (WL+Vest); targeting ≥8 hours/day, weight replacement titrated up to 10% WL); or, WL plus structured RT (WL+RT; 3 days/week). Total hip trabecular volumetric bone mineral density (vBMD) is the primary outcome. This outcome will be complemented by exploratory assessment of several fracture-related risk factors, including: (1) femoral neck and lumbar spine vBMD, cortical thickness, finite element modeling of bone strength, and regional fat and muscle volumes, measured by CT; (2) areal bone mineral density (aBMD) at the total hip, femoral neck, lumbar spine, and distal radius; trabecular bone score; and total body fat/lean masses, measured by dual energy x-ray absorptiometry (DXA); (3) muscle function and strength; (4) biomarkers of bone turnover; and (5) bone-regulating hormones/cytokines known to influence bone metabolism during WL. Therefore, the investigators Specific Aims are to:

Aim 1: Determine the effects of WL+Vest compared to WL and WL+RT on 12 month change in total hip trabecular vBMD. Despite similar reductions in total body weight, Hypothesis 1: Participants in the WL+Vest group will show attenuated losses of total hip trabecular vBMD versus WL; and Hypothesis 2: Loss in total hip trabecular vBMD will be no greater in WL+Vest compared to WL+RT.

Aim 2: Explore the effects of WL+Vest compared to WL and WL+RT on the 12 month change in fracture-related risk factors. Despite similar reductions in total body weight, we hypothesize that WL+Vest and WL+RT will demonstrate improvements in fracture-related risk factors compared to WL.

ELIGIBILITY:
Inclusion Criteria:

* Age 60-85 years
* BMI=30-40 kg/m^2 or BMI 27.0-<30.0 kg/m^2 plus one risk factor
* Weight stability - no weight loss > 5% in past 6 months
* No contraindications for safe and optimal participation in exercise training/vest use.
* Approved for participation by Study Coordinator
* Willing to provide informed consent; agree to all study procedures and assessments; Able to provide own transit to assessment/intervention visits
* Willing to complete online/electronic study forms and participate in virtual group sessions, as needed.

Exclusion Criteria:

* Weight greater than 450 lbs
* Dependent on cane or walker: >2 falls (injurious on non-injurious) in past year
* Any contraindications for participation in voluntary weight loss
* Smoker (>1 cigarette/d or 4/wk within yr); Excessive alcohol use (>14 drinks/wk)
* Participation in regular resistance training and/or high intensity/high impact aerobic exercise for >60 mins per day on > 5 days/week for the past 6 months
* Evidence of cognitive impairment (MoCA<20)
* Osteoporosis (self-report and on prescription medication, T-score < or = -2.5 on total hip, femoral neck, lumbar spine or distal radius scan at screening visit, or fracture risk assessment tool (FRAX) 10-year risk scores >3% for hip fracture or >20% for major osteoporotic fracture (TBS adjusted FRAX is preferable if available)
* Self-reported prior spine, hip, wrist, or shoulder fracture after age 40 (except when caused by trauma or fall from height)
* Chronic back/shoulder/knee pain with current or past (within 1 year) prescription medication use for at least 3 months
* Severe, diagnosed arthritis (osteoarthritis, rheumatoid arthritis, or gout) with current or past (within 1 year) prescription medication use for at least 3 months
* Past (ever) or planned (next 12 months) back surgery
* Past (6 months prior) or planned (next 12 months) joint replacement surgery; or past (ever) unilateral or bilateral hip replacement surgery
* Past (ever) metal device or fixation in the hip, pelvis, or femur
* Uncontrolled hypertension (BP > 160/90 mmHg)
* Current or recent past (within 1 year) severe symptomatic heart disease, uncontrolled angina, stroke, chronic respiratory disease requiring oxygen, neurological or hematological disease requiring treatment for at least 3 months in past year
* Cancer requiring treatment in past year, except non-melanoma skin cancer
* Low Vitamin D (<20 ng/mL)
* Abnormal kidney or liver function (2x upper limits of normal)
* estimated glomerular filtration rate (eGFR)<45 mL/min/1.73m2,
* Anemia (Hb <13 g/dL in men/<12 g/dL in women)
* Uncontrolled diabetes (fasting glucose > 140 mg/dL)
* Regular use of: growth hormones, weight loss medications, oral steroids, insulin, or prescription osteoporosis medications in the past year
* No home computer, laptop or tablet with reliable home internet OR no smartphone (touch-screen enabled phone) with reliable unlimited mobile internet
* Involved in another behavioral/interventional research study, weight loss program, or undergoing physical therapy.
* Unable to tolerate diet, vest, or CT scan (claustrophobia)
* Judged unsuitable for the trial for any reason by clinic staff

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Beavers, PhD, MPH, RD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University School of Medicine, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Beavers KM, Lynch SD, Fanning J, Howard M, Lawrence E, Lenchik L, Shapses SA, Weaver AA, Wherry SJ, Zamora Z, Nicklas BJ, Beavers DP. Weighted Vest Use or Resistance Exercise to Offset Weight Loss-Associated Bone Loss in Older Adults: A Randomized Clinical Trial. JAMA Netw Open. 2025 Jun 2;8(6):e2516772. doi: 10.1001/jamanetworkopen.2025.16772. PMID 40540267
- [Derived] Beavers KM, Avery AE, Shankaran M, Evans WJ, Lynch SD, Dwyer C, Howard M, Beavers DP, Weaver AA, Lenchik L, Cawthon PM. Application of the D3 -creatine muscle mass assessment tool to a geriatric weight loss trial: A pilot study. J Cachexia Sarcopenia Muscle. 2023 Oct;14(5):2350-2358. doi: 10.1002/jcsm.13322. Epub 2023 Sep 5. PMID 37668075
- [Derived] Miller RM, Beavers DP, Cawthon PM, Crotts C, Fanning J, Gerosa J, Greene KA, Hsieh KL, Kiel J, Lawrence E, Lenchik L, Lynch SD, Nesbit BA, Nicklas BJ, Weaver AA, Beavers KM. Incorporating Nutrition, Vests, Education, and Strength Training (INVEST) in Bone Health: Trial Design and Methods. Contemp Clin Trials. 2021 May;104:106326. doi: 10.1016/j.cct.2021.106326. Epub 2021 Feb 22. PMID 33631359

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Weight Loss Plus Vest | Weight Loss Plus Resistance Exercise Training | Weight Loss
Started | 50 | 50 | 50
Completed | 45 | 45 | 43
Not Completed | 5 | 5 | 7
Not completed — Lost to Follow-up | 2 | 1 | 3
Not completed — Withdrawal by Subject | 3 | 1 | 2
Not completed — Relocated out of state | 0 | 2 | 0
Not completed — COVID concerns | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Weight Loss Plus Vest | Weight Loss Plus Resistance Exercise Training | Weight Loss | Total
Number analyzed (Participants) | 50 | 50 | 50 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.9 (4.5) | 66.4 (5.1) | 65.9 (4.2) | 66.4 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 38 | 37 | 112
  Male | 13 | 12 | 13 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 3
  Not Hispanic or Latino | 49 | 49 | 49 | 147
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 16 | 15 | 12 | 43
  White | 33 | 35 | 35 | 103
  More than one race | 1 | 0 | 3 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0
Body Mass Index (kg/m2) [Mean (Standard Deviation); unit: Kilograms] | 93.6 (12.3) | 92.7 (11.9) | 92.3 (14.3) | 92.9 (12.8)
Height [Mean (Standard Deviation); unit: Centimeters] | 166.5 (8.5) | 166.0 (8.0) | 166.0 (8.8) | 166.2 (8.4)
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 33.8 (3.7) | 33.6 (3.0) | 33.4 (3.3) | 33.6 (3.3)
Education [Count of Participants; unit: Participants]
  High School Equivalent | 13 | 7 | 8 | 28
  College | 23 | 27 | 31 | 81
  Post Graduate | 14 | 16 | 11 | 41
Comorbidities [Count of Participants; unit: Participants]
  Diabetes | 5 | 1 | 6 | 12
  Cardiovascular Disease | 4 | 6 | 6 | 16
  Arthritis/Joint Pain | 39 | 29 | 36 | 104
Low Bone Mass [Count of Participants; unit: Participants] | 24 | 23 | 26 | 73
Total Physical Activity [Median (Inter-Quartile Range); unit: Kilocalories Per Week] | 1941 [1272 to 2886] | 2144 [1147 to 3514] | 2042 [1179 to 3345] | 2029 [1179 to 3263]
Fast Gait Speed [Mean (Standard Deviation); unit: Meters Per Second] — Population: 3 participants in the Weight Loss Plus Vest arm did not complete this task at baseline. 2 participants in the Resistance Exercise Training arm did not complete this task at baseline.
  Meters Per Second
    number analyzed (Participants) | 47 | 48 | 50 | 145
    (all) | 1.3 (0.2) | 1.3 (0.2) | 1.3 (0.1) | 1.3 (0.2)
Moderate Intensity Physical Activity [Median (Inter-Quartile Range); unit: Minutes Per Week] | 30 [0 to 165] | 45 [0 to 135] | 0 [0 to 105] | 30 [0 to 135]

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Hip Trabecular Volumetric Bone Mineral Density (vBMD)
Description: measured in mg/cm3 during computed tomography (CT) scan
Time Frame: 12 months from baseline
Population: 6 participants in Weight Loss Plus Vest arm did not complete a CT scan. 5 participants in Weight Loss Plus Resistance Exercise Training arm did not complete a scan. 7 participants in Weight Loss arm did not complete scan.
Measure: Mean (95% Confidence Interval); unit: mg/cm3
Arm/Group | Weight Loss Plus Vest | Weight Loss Plus Resistance Exercise Training | Weight Loss
Number analyzed (Participants) | 44 | 45 | 43
mg/cm3 | -0.002 [-0.003 to -0.001] | -0.002 [-0.003 to -0.001] | -0.003 [-0.003 to -0.002]

2. Secondary Outcome: Change in Total Hip Trabecular Volumetric Bone Mineral Density (vBMD)
Description: measured in mg/cm3 during computed tomography (CT) scan
Time Frame: 6 months from baseline
Population: 4 participants in Weight Loss Plus Vest arm did not complete a CT scan. 4 participants in Weight Loss Plus Resistance Exercise Training arm did not complete a scan. 6 participants in Weight Loss arm did not complete scan.
Measure: Mean (95% Confidence Interval); unit: mg/cm3
Arm/Group | Weight Loss Plus Vest | Weight Loss Plus Resistance Exercise Training | Weight Loss
Number analyzed (Participants) | 46 | 46 | 44
mg/cm3 | -0.001 [-0.001 to 0.000] | -0.000 [-0.001 to 0.001] | -0.000 [-0.001 to 0.000]

3. Secondary Outcome: Change in Femoral Neck Volumetric Bone Mineral Density (vBMD)
Description: measured in mg/cm3 during computed tomography (CT) scan
Time Frame: 6 months from baseline
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: mg/cm3
Arm/Group | Weight Loss Plus Vest | Weight Loss Plus Resistance Exercise Training | Weight Loss
Number analyzed (Participants) | 46 | 46 | 44
mg/cm3 | -0.001 [-0.003 to 0.001] | -0.001 [-0.003 to 0.001] | -0.001 [-0.002 to 0.001]

4. Secondary Outcome: Change in Femoral Neck Volumetric Bone Mineral Density (vBMD)
Description: measured in mg/cm3 during computed tomography (CT) scan
Time Frame: 12 months from baseline
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mg/cm3
Arm/Group | Weight Loss Plus Vest | Weight Loss Plus Resistance Exercise Training | Weight Loss
Number analyzed (Participants) | 44 | 45 | 43
mg/cm3 | -0.002 [-0.004 to 0.001] | -0.003 [-0.005 to -0.000] | -0.004 [-0.007 to -0.002]

5. Secondary Outcome: Change in Lumbar Spine Volumetric Bone Mineral Density (vBMD)
Description: measured in mg/cm3 during computed tomography (CT) scan
Time Frame: 6 months from baseline
Population: 3 participants in Weight Loss Plus Vest arm did not complete the scan. 4 participants in Weight Loss Plus Resistance Exercise Training arm did not complete the scan. 5 participants in the Weight Loss arm did not complete the scan.
Measure: Mean (95% Confidence Interval); unit: mg/cm3
Arm/Group | Weight Loss Plus Vest | Weight Loss Plus Resistance Exercise Training | Weight Loss
Number analyzed (Participants) | 47 | 46 | 45
mg/cm3 | 0.001 [-0.002 to 0.005] | 0.005 [0.001 to 0.008] | 0.005 [0.002 to 0.008]

6. Secondary Outcome: Change in Lumbar Spine Volumetric Bone Mineral Density (vBMD)
Description: measured in mg/cm3 during computed tomography (CT) scan
Time Frame: 12 months from baseline
Population: 5 participants in Weight Loss Plus Vest arm did not complete the scan. 5 participants in Weight Loss Plus Resistance Exercise Training arm did not complete the scan. 7 participants in the Weight Loss arm did not complete the scan.
Measure: Mean (95% Confidence Interval); unit: mg/cm3
Arm/Group | Weight Loss Plus Vest | Weight Loss Plus Resistance Exercise Training | Weight Loss
Number analyzed (Participants) | 45 | 45 | 43
mg/cm3 | -0.000 [-0.002 to 0.002] | 0.003 [0.001 to 0.005] | 0.000 [-0.002 to 0.002]

7. Secondary Outcome: Change in Trabecular Bone Score (TBS)
Description: measurement taken during dual energy x-ray absorptiometry (DXA) scan; Trabecular Bone Score is a measure of bone architecture that has been shown to be an independent risk factor for fracture. The measure is unitless, and ranges from 1.0-1.6, where an elevated TBS greater than or equal to 1.3 appears to represent strong, fracture-resistant bone architecture, while a low TBS less than or equal to 1.2 reflects weak, fracture-prone bone architecture.
Time Frame: 6 months from baseline
Population: 3 participants in Weight Loss Plus Vest arm did not complete DXA scan. 3 participants in Weight Loss Plus Resistance Exercise Training Arm did not complete DXA scan. 5 participants in Weight Loss arm did not complete DXA scan.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Weight Loss Plus Vest | Weight Loss Plus Resistance Exercise Training | Weight Loss
Number analyzed (Participants) | 47 | 47 | 45
score on a scale | 0.020 [0.002 to 0.039] | 0.037 [0.018 to 0.056] | 0.017 [-0.002 to 0.035]

8. Secondary Outcome: Change in Trabecular Bone Score (TBS)
Description: as for outcome 7
Time Frame: 12 months from baseline
Population: 5 participants in Weight Loss Plus Vest arm did not complete DXA scan. 5 participants in Weight Loss Plus Resistance Exercise Training Arm did not complete DXA scan. 7 participants in Weight Loss arm did not complete DXA scan.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Weight Loss Plus Vest | Weight Loss Plus Resistance Exercise Training | Weight Loss
Number analyzed (Participants) | 45 | 45 | 43
score on a scale | 0.014 [-0.005 to 0.034] | 0.037 [0.017 to 0.057] | 0.017 [-0.003 to 0.037]

9. Secondary Outcome: Change in Total Hip Areal Bone Mineral Density (aBMD)
Description: measured in g/cm2 during dual energy x-ray absorptiometry (DXA) scan
Time Frame: 6 months from baseline
Population: 3 participants in Weight Loss Plus Vest did not complete DXA scan. 3 participants in Weight Loss Plus Resistance Exercise Training arm did not complete DXA scan. 5 participants in Weight Loss arm did not complete DXA scan.
Measure: Mean (95% Confidence Interval); unit: g/cm2
Arm/Group | Weight Loss Plus Vest | Weight Loss Plus Resistance Exercise Training | Weight Loss
Number analyzed (Participants) | 47 | 47 | 45
g/cm2 | -0.006 [-0.013 to 0.001] | -0.008 [-0.015 to -0.001] | -0.008 [-0.015 to -0.001]

10. Secondary Outcome: Change in Total Hip Areal Bone Mineral Density (aBMD)
Description: measured in g/cm2 during dual energy x-ray absorptiometry (DXA) scan
Time Frame: 12 months from baseline
Population: 5 participants in Weight Loss Plus Vest did not complete DXA scan. 5 participants in Weight Loss Plus Resistance Exercise Training arm did not complete DXA scan. 7 participants in Weight Loss arm did not complete DXA scan.
Measure: Mean (95% Confidence Interval); unit: g/cm2
Arm/Group | Weight Loss Plus Vest | Weight Loss Plus Resistance Exercise Training | Weight Loss
Number analyzed (Participants) | 45 | 45 | 43
g/cm2 | -0.015 [-0.023 to -0.007] | -0.016 [-0.024 to -0.008] | -0.017 [-0.025 to -0.009]

11. Secondary Outcome: Change in Femoral Neck Areal Bone Mineral Density (aBMD)
Description: measured in g/cm2 during dual energy x-ray absorptiometry (DXA) scan
Time Frame: 6 months from baseline
Population: as for outcome 7
Measure: Mean (95% Confidence Interval); unit: g/cm2
Arm/Group | Weight Loss Plus Vest | Weight Loss Plus Resistance Exercise Training | Weight Loss
Number analyzed (Participants) | 47 | 47 | 45
g/cm2 | -0.000 [-0.011 to 0.010] | 0.004 [-0.007 to 0.014] | 0.004 [-0.007 to 0.015]

12. Secondary Outcome: Change in Femoral Neck Areal Bone Mineral Density (aBMD)
Description: measured in g/cm2 during dual energy x-ray absorptiometry (DXA) scan
Time Frame: 12 months from baseline
Population: as for outcome 8
Measure: Mean (95% Confidence Interval); unit: g/cm2
Arm/Group | Weight Loss Plus Vest | Weight Loss Plus Resistance Exercise Training | Weight Loss
Number analyzed (Participants) | 45 | 45 | 43
g/cm2 | -0.006 [-0.017 to 0.005] | -0.004 [-0.015 to 0.008] | -0.005 [-0.016 to 0.007]

13. Secondary Outcome: Change in Distal Radius Areal Bone Mineral Density (aBMD)
Description: measured in g/cm2 during dual energy x-ray absorptiometry (DXA) scan
Time Frame: 6 months from baseline
Population: 3 participants in the Weight Loss Plus Vest arm did not complete DXA scan. 3 participants in the Weight Loss Plus Resistance Exercise Training arm did not complete DXA scan. 5 participants in the Weight Loss arm did not complete DXA scan.
Measure: Mean (95% Confidence Interval); unit: g/cm2
Arm/Group | Weight Loss Plus Vest | Weight Loss Plus Resistance Exercise Training | Weight Loss
Number analyzed (Participants) | 47 | 47 | 45
g/cm2 | -0.009 [-0.018 to 0.000] | -0.008 [-0.018 to 0.001] | -0.007 [-0.016 to 0.002]

14. Secondary Outcome: Change in Distal Radius Areal Bone Mineral Density (aBMD)
Description: measured in g/cm2 during dual energy x-ray absorptiometry (DXA) scan
Time Frame: 12 months from baseline
Population: 5 participants in the Weight Loss Plus Vest arm did not complete DXA scan. 5 participants in the Weight Loss Plus Resistance Exercise Training arm did not complete DXA scan. 7 participants in the Weight Loss arm did not complete DXA scan.
Measure: Mean (95% Confidence Interval); unit: g/cm2
Arm/Group | Weight Loss Plus Vest | Weight Loss Plus Resistance Exercise Training | Weight Loss
Number analyzed (Participants) | 45 | 45 | 43
g/cm2 | -0.013 [-0.022 to -0.003] | -0.007 [-0.017 to 0.003] | -0.013 [-0.022 to -0.003]

15. Secondary Outcome: Change in Lumbar Spine Areal Bone Mineral Density (aBMD)
Description: measured in g/cm2 during dual energy x-ray absorptiometry (DXA) scan
Time Frame: 6 months from baseline
Population: as for outcome 7
Measure: Mean (95% Confidence Interval); unit: g/cm2
Arm/Group | Weight Loss Plus Vest | Weight Loss Plus Resistance Exercise Training | Weight Loss
Number analyzed (Participants) | 47 | 47 | 45
g/cm2 | 0.003 [-0.011 to 0.017] | 0.015 [0.000 to 0.030] | 0.016 [0.001 to 0.030]

16. Secondary Outcome: Change in Lumbar Spine Areal Bone Mineral Density (aBMD)
Description: measured in g/cm2 during dual energy x-ray absorptiometry (DXA) scan
Time Frame: 12 months from baseline
Population: as for outcome 8
Measure: Mean (95% Confidence Interval); unit: g/cm2
Arm/Group | Weight Loss Plus Vest | Weight Loss Plus Resistance Exercise Training | Weight Loss
Number analyzed (Participants) | 45 | 45 | 43
g/cm2 | 0.006 [-0.012 to 0.023] | 0.011 [-0.007 to 0.028] | 0.010 [-0.008 to 0.027]

17. Secondary Outcome: Change in Total Body Fat Mass (kg)
Description: measurement taken during dual energy x-ray absorptiometry (DXA) scan
Time Frame: 6 months from baseline
Population: as for outcome 7
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Weight Loss Plus Vest | Weight Loss Plus Resistance Exercise Training | Weight Loss
Number analyzed (Participants) | 47 | 47 | 45
kg | -7.8 [-9.1 to -6.5] | -8.8 [-10.2 to -7.5] | -7.8 [-9.2 to -6.5]

18. Secondary Outcome: Change in Total Body Fat Mass (kg)
Description: measurement taken during dual energy x-ray absorptiometry (DXA) scan
Time Frame: 12 months from baseline
Population: as for outcome 8
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Weight Loss Plus Vest | Weight Loss Plus Resistance Exercise Training | Weight Loss
Number analyzed (Participants) | 45 | 45 | 43
kg | -7.3 [-8.9 to -5.7] | -10.0 [-11.6 to -8.3] | -7.7 [-9.4 to -6.0]

19. Secondary Outcome: Change in Total Body Lean Mass (kg)
Description: measurement taken during dual energy x-ray absorptiometry (DXA)
Time Frame: 6 months from baseline
Population: as for outcome 7
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Weight Loss Plus Vest | Weight Loss Plus Resistance Exercise Training | Weight Loss
Number analyzed (Participants) | 47 | 47 | 45
kg | -0.5 [-1.1 to 0.0] | -0.8 [-1.4 to -0.2] | -0.7 [-1.2 to -0.1]

20. Secondary Outcome: Change in Total Body Lean Mass (kg)
Description: measurement taken during dual energy x-ray absorptiometry (DXA)
Time Frame: 12 months from baseline
Population: as for outcome 8
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Weight Loss Plus Vest | Weight Loss Plus Resistance Exercise Training | Weight Loss
Number analyzed (Participants) | 45 | 45 | 43
kg | -0.7 [-1.3 to -0.2] | -0.9 [-1.4 to -0.3] | -0.9 [-1.5 to -0.4]

21. Other Pre Specified Outcome: Mid-thigh Muscle Density Measured in Hounsfield Units (HU)
Description: measurement taken during computed tomography (CT) scan
Time Frame: 12 months from baseline
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Mid- Thigh Intermuscular Fat Cross Sectional Area (CSA) (cm2)
Description: measurement taken during computed tomography (CT) scan
Time Frame: 12 months from baseline
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Cortical Thickness (mm)
Description: measurement taken during computed tomography (CT) scan
Time Frame: 12 months from baseline
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Finite Element (FE) Modeling of Bone Strength Measured in Kilonewton (kN)
Description: measurement taken during computed tomography (CT) scan
Time Frame: 12 months from baseline
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Mid-thigh Muscle CSA (cm2)
Description: measurement taken during computed tomography (CT) scan
Time Frame: 12 months from baseline
Reporting Status: Not Posted

26. Other Pre Specified Outcome: L3 Muscle Density Measured in HU
Description: measurement taken during computed tomography (CT) scan
Time Frame: 12 months from baseline
Reporting Status: Not Posted

27. Other Pre Specified Outcome: L3 Intermuscular Fat CSA (cm2)
Description: measurement taken during computed tomography (CT) scan
Time Frame: 12 months from baseline
Reporting Status: Not Posted

28. Other Pre Specified Outcome: L3 Muscle CSA (cm2)
Description: measurement taken during computed tomography (CT) scan
Time Frame: 12 months from baseline
Reporting Status: Not Posted

29. Other Pre Specified Outcome: Concentration of Procollagen 1 Intact N-Terminal Propeptide (P1NP) (ug/L)
Description: Biomarkers of bone turnover measured via blood specimen
Time Frame: 12 months from baseline
Reporting Status: Not Posted

30. Other Pre Specified Outcome: Concentration of C-terminal Telopeptide (CTX) (pg/mL)
Description: Biomarkers of bone turnover measured via blood specimen
Time Frame: 12 months from baseline
Reporting Status: Not Posted

31. Other Pre Specified Outcome: D3-Creatine Derived Muscle Mass Measured in kg
Description: measurement taken via urine sample
Time Frame: 12 months from baseline
Reporting Status: Not Posted

32. Other Pre Specified Outcome: Gait Speed
Description: measured in m/s during the 400 meter walk test
Time Frame: 12 months from baseline
Reporting Status: Not Posted

33. Other Pre Specified Outcome: Expanded Short Physical Performance Battery (eSPPB)
Description: The SPPB is a measure of balance, walking speed, and ability to stand from a chair. It provides a global measure of overall physical function and is a good predictor of future disability, institutionalization, and mortality in older persons. The SPPB score is calculated by assigning each of the test measures (balance, walking speed, and chair stands) a score from 0 (unable to do) to 4 (best) and then adding these scores together for a total score ranging from 0 to 12. An SPPB score less than 10 identifies persons at higher risk for mobility disability.
Time Frame: 12 months from baseline
Reporting Status: Not Posted

34. Other Pre Specified Outcome: Timed-Up-and-Go (TUG)
Description: measured in seconds to assess physical performance; measures the time the participant takes to stand up from a standard chair, walk 3 meters, turn, walk back to the chair, and sit down again.
Time Frame: 12 months from baseline
Reporting Status: Not Posted

35. Other Pre Specified Outcome: Stair Climbing Time
Description: measured in seconds using the participant's fastest time achieved to climb a 12 step staircase in two trials.
Time Frame: 12 months from baseline
Reporting Status: Not Posted

36. Other Pre Specified Outcome: Lower Extremity Muscle Strength
Description: measured using an isokinetic dynamometer with the participant sitting and the hips and knee flexed at 90°. Participants will be asked to extend the knee and push as hard as possible against the resistance pad. Strength is expressed as peak torque (Nm)
Time Frame: 12 months from baseline
Reporting Status: Not Posted

37. Other Pre Specified Outcome: Grip Strength
Description: measured twice in each hand to the nearest two kg using an isometric Jamar Hydraulic Hand Dynamometer with the mean value from the stronger hand used
Time Frame: 12 months from baseline
Reporting Status: Not Posted

38. Other Pre Specified Outcome: Cognitive Assessment
Description: measured using the Montreal Cognitive Assessment (MOCA) with scores ranging from 0-30, with a score of 26 and higher generally considered normal.
Time Frame: 12 months from baseline
Reporting Status: Not Posted

39. Other Pre Specified Outcome: Fatigability
Description: measured using the Pittsburgh Fatigability scale, which is a 10-item questionnaire that assesses fatigability, or the rate at which a person experiences mental or physical fatigue in the context of a standardized task. The scale ranges from 0-5, where those who exhibit more fatigability, score of 5, are more likely to limit activities of daily living and to reduce exertion during physical activities.
Time Frame: 12 months from baseline
Reporting Status: Not Posted

40. Other Pre Specified Outcome: Pain and Fatigue
Description: measured using The Patient-Reported Outcomes Measurement Information System (PROMIS) instrument is an 8-item short-form that assesses pain and fatigue over the past 7 days. The scale ranges from 1-5, with higher scores indicated the presence of pain and fatigue.
Time Frame: 12 months from baseline
Reporting Status: Not Posted

41. Other Pre Specified Outcome: Physical Activity Among Older Adults
Description: The CHAMPS questionnaire is a 40-43-item tool that assesses weekly frequency and duration of a variety of lifestyle physical activities that are appropriate for older adults. The purpose of this questionnaire is to evaluate the effectiveness of interventions to increase lifestyle physical activity among older adults. Physical activities are given a METS score, ranging from 2.0-7.0, where activities with an activities of moderate intensity (METS) score of 3.0 or higher, are considered moderate intensity.
Time Frame: 12 months from baseline
Reporting Status: Not Posted

42. Other Pre Specified Outcome: Overall Limb Loading
Description: measured in Newtons via force-sensing insoles to assess overall limb loading and to determine if participants receive enough loading to prevent bone loss from resistance training and weighted vest use when compared to weight loss alone.
Time Frame: 6 months from baseline
Reporting Status: Not Posted

43. Other Pre Specified Outcome: Overall Satisfaction Participating in the Optional Insole Visits
Description: overall satisfaction measured by a scale from 1-5 with a higher score indicating greater satisfaction
Time Frame: 6 months from baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Baseline through Month 12
Arm/Group | Weight Loss Plus Vest | Weight Loss Plus Resistance Exercise Training | Weight Loss
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 3/50 | 1/50 | 2/50
Other Adverse Events (participants affected / at risk) | 23/50 | 22/50 | 20/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Weight Loss Plus Vest (N=50) | Weight Loss Plus Resistance Exercise Training (N=50) | Weight Loss (N=50)
Small bowel obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Motor vehicle accident (Social circumstances) | 1 (1) | 0 (0) | 0 (0)
Prostate transurethral resection (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Weight Loss Plus Vest (N=50) | Weight Loss Plus Resistance Exercise Training (N=50) | Weight Loss (N=50)
Fall (Social circumstances) | 12 (14) | 6 (7) | 10 (10)
COVID-19 (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 10 (11) | 5 (5)
Sinusitis (Infections and infestations) | 2 (2) | 2 (2) | 6 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 3 (3) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 2 (2) | 3 (4) | 1 (1)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 1 (1)
Knee pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-04): https://cdn.clinicaltrials.gov/large-docs/18/NCT04076618/Prot_SAP_001.pdf
  • Informed Consent Form (2024-03-05): https://cdn.clinicaltrials.gov/large-docs/18/NCT04076618/ICF_000.pdf